CLINICAL TRIAL: NCT04865549
Title: Sentinel Node After Neoadjuvancy In Node-Positive Breast Cancer: SANA Multicentric Study
Brief Title: Sentinel Node After Neoadjuvancy In Node-Positive Breast Cancer
Acronym: SANA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HCB/2016/0296
Record Dates: First submitted 2021-04-12; First posted 2021-04-29 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — DAT protocol 1; Lymph Node Excision

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TAD arm (Experimental): Sentinel Node Biopsy + Targetted Axillary Dissection (Clipped cN1 node) extraction + lymphadenectomy.
  Interventions: Procedure: SNB + TAD + Lymphadenectomy

INTERVENTIONS:
Procedure: SNB + TAD + Lymphadenectomy — Sentinel Node Biopsy + Targetted Axillary Dissection (Previously to surgery marked cN1 node) + Lymphadenectomy

SUMMARY:
The status of the axillary lymph nodes is one of the main prognostic factors in breast cancer (BC). SLNB is currently the standard staging method for patients with clinically node-negative (cN0) breast cancer. In patients with a positive SLN and in those with affected lymph nodes at the beginning (cN+), LND is the standard of treatment.

DETAILED DESCRIPTION:
Breast cancer (BC) is the most common malignant tumor and the one that causes the highest number of deaths among women around the world. In Spain some 25,000 new cases are diagnosed per year, which represents almost 30% of all female tumors. In Catalonia, the incidence is 83.9 cases / 100,000 inhabitants, while the national average is 50.9 cases / 100,000 inhabitants.

Thanks to screening programs and the awareness of patients and professionals, the majority of diagnosed cases are found in an early stage of the disease. In early stages, the prognosis is excellent with a 5-year survival greater than 80%.

Lymph node staging: selective sentinel node biopsy (SLNB) vs axillary lymphadenectomy The status of the axillary lymph nodes is one of the main prognostic factors. Knowing the lymph node status allows the disease to be staged and modulates locoregional and systemic treatment. Lymph node staging and management of axillary disease have changed dramatically in recent decades.

SLNB is currently the standard staging method for patients with clinically node-negative (cN0) breast cancer. When SLN is negative, axillary lymph node dissection (LND) can be omitted without prejudice to patient survival or locoregional control of the disease. In patients with a positive SLN and in those with affected lymph nodes at the beginning (cN+), LND is the standard of treatment. Morbidity associated with this technique affects up to 80% of patients and includes: chronic lymphedema of the upper limb (20-30%), seromas (50-60%) that in many cases require repeated punctures for drainage, infection of the wound (5-15%) that requires antibiotic treatment and sometimes drainage, decreased mobility of the arm or "frozen shoulder" (up to 10%) that requires rehabilitation treatment, neuropathic pain due to injury to the intercostobrachial nerve (5- 20%) and other less frequent ones such as hematoma or section of the long thoracic nerves (which produces a scapula alata) or the latissimus dorsi. It is obvious that all these complications affect the quality of life of patients and their emotional state. LND lengthens the days of hospitalization and this, together with the treatment of associated complications, substantially increases healthcare costs.

Current focus on the initial treatment of breast cancer: primary systemic treatment Advances in biological knowledge of the disease and in systemic treatments have led to an increasing number of patients with BC starting with systemic therapy, relegating surgery to a second stage. This approach evaluates the tumor response in vivo to systemic treatment and provides critical prognostic information. In addition, the decrease and even disappearance of the tumor increases the chances of offering a conservative surgery in the breast. Response rates vary according to the biological type of tumor and the treatment used, being higher for Her2+ tumors treated with chemotherapy combined with anti-Her2 antibodies.

In cN0 patients receiving neoadjuvant chemotherapy (NCT), SLNB can be performed before or after. Performing it later, together with breast surgery, has the advantage of saving the patient a surgical procedure. This strategy is supported by numerous studies that show detection and false negative (FN) rates comparable to those of patients who undergo SLNB before neoadjuvant treatment.

In those patients who present clinically positive lymph nodes (cN +) before initiating neoadjuvancy, the standard strategy in relation to the axilla is to perform LND. However, in 40-50% of patients, lymph node disease disappears with treatment. Nodal response is greater in tumors with estrogen receptor negative, high histologic grade, and Her2 overexpression. It follows that up to 40-50% of unnecessary lymphadenectomies are currently being carried out.

Application of the SLNB in cN + patients undergoing neoadjuvant chemotherapy Due to the benefits that SLNB represents in cN0 patients and the complete response rates in the axilla after neoadjuvant chemotherapy (NAC) in initial cN+ patients, the question arises as to whether SLNB can be valid in these patients. Previous studies in which SLNB was performed in clinically node-positive patients who received NAC have shown FN rates of up to 25%. The Spanish Society of Senology and Breast Pathology (SESPM) recommends for the validation of the SLN technique to obtain a detection rate equal to or greater than 95% and a FN rate equal to or less than 5%. International literature accepts FN rates equal to or less than 10%.

The success of SLNB after NAC may be affected by altered lymphatic drainage of the breast during chemotherapy. On the other hand, it is possible that the regression of the axillary disease does not follow an orderly and uniform pattern, reducing the reliability of the technique. Finally, the impact that a FN of the technique may have on the prognosis of these patients is unknown, and it is probably not the same as in a cN0 patient.

The American College of Surgeons Oncology Group (ACOSOG) conducted a phase II trial that included patients with BC T1-4, N1-2, M0. The patients received primary chemotherapy and subsequently SLNB plus LND. The detection rate was 92.9%. There was a complete pathological response in the axilla in 41% of the patients. The FN rate was 12.6% (higher than the accepted 10%). The conclusion was that SLN biopsy cannot be recommended for these patients at this time.

The multicenter study SENTINA (SENTinel NeoAdjuvant), carried out in Germany and Austria, evaluated in one of its arms the performance of SLNB in cN + patients who converted to cN0 with NAC. The SLN detection rate and the FN rate were 80.1% and 14.2%, respectively. None of these studies evaluate the results of the technique based on the biological profile of the tumor or the response of the disease to treatment.

It is imperative to correctly select patients and apply new strategies to optimize the results of SLNB in order to identify regression of axillary disease and to avoid radicality of LA.

New strategies: placement of a marker in the metastatic lymph node. Assessment of the response according to the biological profile of the tumor and its impact on the rate of FN Axillary ultrasound prior to neoadjuvancy is performed to detect possible lymph node involvement and, together with biopsy of the suspicious node, offers a sensitivity and specificity of 25% -95% and 97% -100%, respectively. Its application could be useful to assess axillary lymph node response. Patients with normal-appearing axillary nodes on ultrasound are likely to be less likely to have residual disease.

The placement of a marker in the biopsied pathological node that allows its identification during the surgical act and to check whether or not it correlates with the SLN can be useful strategies to reduce the rate of FN of the SLNB.

The response of the disease in the breast and in the lymph nodes to NAC is different depending on the biological profile of the tumor. The axillary response to treatment may have an impact on the rate of FN of SLNB. Studying the results of the technique according to the biological profile of the tumor can help us to better select the candidate patients for the application of the technique.

ELIGIBILITY:
Inclusion Criteria:

* Age equal to or greater than 18 years
* Patients with a diagnosis of T1-T3 primary infiltrating breast carcinoma
* Axillary clinical involvement (cN +)
* Confirmation by FNAC or BAG of lymph node involvement
* Candidates for neoadjuvant chemotherapy including anthracyclines and taxanes

Exclusion Criteria:

* T4 tumors
* Supra / infraclavicular lymph node or internal mammary chain (cN3) involvement
* Previous ipsilateral breast or axillary surgery
* Distant metastasis at diagnosis (M1)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Targetted axilary dissection detection rate in cN+ after neoadjuvant therapy | immediately after surgery
  Targetted axilary dissection detection rate in cN+ after neoadjuvant therapy (Sentinel lymph node plus cliped node)

SECONDARY OUTCOMES:
False negative Rate | immediately after surgery
  To know the detection rate and the false negative rate of the SLN biopsy in cN + patients.
Concordance | immediately after surgery
  Know the concordance rate between the SLN and the pathological node marked with an echo-visible marker
Ultrasound before-after NAC | before the start of systemic therapy - after finishing systemic therapy just before surgery
  To study the usefulness of axillary ultrasound before and after NAC to assess lymph node involvement and response to treatment
Response Rate by biological profile | immediately after the intervention/procedure/surgery
  Assess the axillary lymph node response rate based on the biological profile of the tumor
Response Rate by treatment | immediately after the intervention/procedure/surgery
  Assess the axillary lymph node response rate based on the primary systemic treatment received.
Risk factors description | immediately after the intervention/procedure/surgery
  Study factors that influence detection rates and FN: marker placement in the pathological node of origin, method of SN identification; number of GC obtained; systemic treatment received; clinical and radiological response to treatment
False Negative Rate by biological profile | immediately after the intervention/procedure/surgery
  To study specifically the influence of the biological profile of the tumor on the FN rate of the technique

CONTACTS AND LOCATIONS:
Overall Officials: Immaculada Alonso Vargas, MD PhD, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clínic de Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No